CLINICAL TRIAL: NCT02673827
Title: Effect of Progressive Muscle Relaxation as a Nursing Intervention on Sleep Quality, Depression and Stress in People With Multiple Sclerosis
Brief Title: Progressive Muscle Relaxation Effect on Sleep Quality, Depression and Stress in People With Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of Espirito Santo (Other)
Responsible Party: Principal Investigator, Paolla Gabrielle Nascimento Novais, Principal investigator, Federal University of Espirito Santo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 618.841/2014
Record Dates: First submitted 2016-01-28; First posted 2016-02-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Multiple Sclerosis; Depression; Sleep; Stress Psychological
MeSH Terms: conditions — Multiple Sclerosis; Depression; Stress, Psychological | interventions — Autogenic Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group control (No Intervention): Control group: 20 patients with relapsing-remitting multiple sclerosis only receive traditional treatment.
- experimental group (Experimental): Intervention group: 20 patients with relapsing-remitting multiple sclerosis receive five sessions of Progressive Muscle Relaxation under the supervision of a researcher in neurology clinic. Before and after each session of the Progressive Muscle Relaxation.
  They will be measured heart rate, respiratory rate and blood pressure. Participants will be guided to realize the Progressive Muscle Relaxation daily for 8 weeks, the time of day you feel more comfortable. the same receive education and training as the technical as well as a audio and a leaflet with the description the stages of the Progressive Muscle Relaxation.
  Interventions: Other: Progressive muscle relaxation

INTERVENTIONS:
Other: Progressive muscle relaxation — Intervention group: 20 patients with relapsing-remitting multiple sclerosis receive five sessions of Progressive Muscle Relaxation under the supervision of a researcher in neurology clinic. Before and after each session of the Progressive Muscle Relaxation They will be measured heart rate, respiratory rate and blood pressure. Participants will be guided to realize the Progressive Muscle Relaxation daily for 8 weeks, the time of day you feel more comfortable. the same receive education and training as the technical as well as a audio and a leaflet with the description the stages of the Progressive Muscle Relaxation. Control group: 20 patients with relapsing-remitting multiple sclerosis only receive traditional treatment.
  Arms: experimental group

SUMMARY:
Objective: Evaluate the effects of Progressive Muscle Relaxation on sleep quality and on stress and depression levels of individuals with multiple sclerosis.

DETAILED DESCRIPTION:
Introduction: Multiple sclerosis is a chronic, autoimmune disease, characterized by demyelination and neurodegeneration of the central nervous system. The progressive course of this disease may cause individuals to develop extreme dependency and create serious difficulties both to the individuals themselves and family members and caregivers, since the disease brings a number of physical, emotional, psychological and social symptoms. Therefore, it is essential to offer healthcare practices that go beyond the usually fragmenting, dehumanized care services that focus on the disease bodily processes.

Objective: Evaluate the effects of Progressive Muscle Relaxation on sleep quality and on stress and depression levels of individuals with multiple sclerosis.

Methodology: This is randomized clinical test. The sample was made up of 40 individuals with multiple sclerosis (20 in control group and 20 in the experimental group) in outpatient follow-up. The progressive muscle relaxation technique was employed. In order to collect the data, we adopted the interview with form filling technique, using the Pittsburgh Sleep Quality Index, Perceived Stress Scale and Beck Depression Inventory. Blood pressure, heart rate and respiratory rate of experimental group were measured before and after the progressive muscle relaxation intervention. In order to treat statistical data, we used Statistical Package for Social Sciences, version 19.0.

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed with Multiple Sclerosis for at least 6 months
* To be diagnosed with relapsing-remitting multiple sclerosis
* To have Expanded Disability Status Scale score < 5.0
* To not have had any attacks during the 3-month period preceding enrollment in the study
* To have audio at home
* To be residing in the Metropolitan region of Vitória-Espirito Santo-Brazil.
* To be 18-65 years of age
* Treatment with an immunomodulator

Exclusion Criteria:

* Being hospitalized at the time of data collection or outbreak at the time of data collection
* Have physical and / or mental changes that prevent the collection of data, such as motor or cognitive deficits
* Experiencing relapse and/or corticosteroid use within the last month, diagnosed with progressive MS (primary or secondary)
* Use of psychotropic drugs (antidepressants, benzodiazepines, antipsychotic and cannabis, or other stimulants),
* Practice of other relaxation techniques (yoga, pilates, meditation, psychotherapy)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-04; Primary Completion 2014-10 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Stress Level | 2 months
  Instrument: Perceived Stress Scale.

SECONDARY OUTCOMES:
Level of depression | 2 months
  Instrument : Beck Depression Inventory.
sleep quality | 2 months
  Instrument: Pittsburgh Sleep Quality Index.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Novais PG, Batista Kde M, Grazziano Eda S, Amorim MH. The effects of progressive muscular relaxation as a nursing procedure used for those who suffer from stress due to multiple sclerosis. Rev Lat Am Enfermagem. 2016 Sep 1;24:e2789. doi: 10.1590/1518-8345.1257.2789. PMID 27598379